CLINICAL TRIAL: NCT07089394
Title: Retrograde Intrarenal Surgery for Renal Stones in Pediatrics: A Prospective Analysis of Feasibility and Outcomes.
Acronym: RIRS pediatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Emad Gouda, urology assistant lecturer, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7603
Record Dates: First submitted 2025-07-21; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Renal Stones; Pediatric Renal Stones
Keywords: pediatric; renal stones; flexible ureteroscopy; holmium laser
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pediatric patients presented with ≤2cm renal stones within 2 years from jan 2023 to jan 2025 (Other): treatment of pediatric renal stones ≤2cmwith flexible URS +Holmium laser fragmentation
  Interventions: Procedure: flexible urs

INTERVENTIONS:
Procedure: flexible urs — treating pediatric renal stones with flexible urs+holmium laser fragmentation
  Other Names: RIRS; FURS

SUMMARY:
it is an interventional single arm study for treating pediatric renal stones≤2cm by FURS and Holmium laser fragmentation.pediatric groups is benig compared for stone free rate, complication rate , success rate. 3 groups of children . group 1 up to 6 years, group 2 from 7 to 12 years , group 3 from 13 to 18 years

ELIGIBILITY:
Inclusion Criteria:

* pediatric renal stones ≤2cm indicated for treatment

Exclusion Criteria:

* congenital urinary tract anomalies, coagulation disorders, active uti,distal ureteric obstruction, bigger stone size

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
stone free rate | within 2 months after intervention
  stone free rate as proved by ctut ,defined as fragments ≤2 mm fragment

SECONDARY OUTCOMES:
complication rate among all groups | intra, post operative, untill stent removal or within 2 months after intervention
  complication rate over all and in each pediatric group in comparative analysis

CONTACTS AND LOCATIONS:
Locations (1):
- AlAzhar university hospitals/Urology department, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results and publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2025 till 2026

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT07089394/Prot_SAP_000.pdf